CLINICAL TRIAL: NCT01385397
Title: Integrated Obesity Care Management System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Marie-France Langlois, Professor, Université de Sherbrooke
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 05-109
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Obesity
Keywords: Health system organization
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preceptorship and virtual community (Experimental)
  Interventions: Other: Preceptorship and virtual community

INTERVENTIONS:
Other: Preceptorship and virtual community

SUMMARY:
Obesity is an important public health problem that is taking epidemic proportions worldwide. Indeed, nearly 50% of Canadians are obese and their number has increased dramatically in the last 20 years. Direct costs of obesity added to those of sedentary represent nearly 5% of the health system's budget. Also, obesity is linked with multiple co-morbidities; furthermore, modest weight loss has significant impact on type 2 diabetes, blood pressure and even reduces mortality. The investigators group has implemented an interdisciplinary team that has demonstrated its effectiveness for obesity management. However, the majority of obese subjects should be treated by primary care physicians (PCPs) that often feel uncomfortable when faced with the management of obesity. The investigators have therefore developed a clinical preceptorship for PCPs; this continuing medical education (CME) activity aims at engaging PCPs in obesity/overweight management. The current research proposal is aimed at the development and implementation of an innovative, integrated, interdisciplinary obesity care management system involving both primary and secondary health care professionals.

The investigators hypothesize that CME based on preceptorships in combination with electronic tools (web site and virtual community), networking primary care (FMGs) and secondary care health professionals, will increase the knowledge, modify attitudes and perceptions of health care professionals and increase their sense of self-efficacy. Furthermore, this intervention should modify health care organization regarding obesity management and eventually improve accessibility to optimal obesity care.

The investigators will use both action (objectives 1-2) and evaluative (objectives 3-5) research in order to attain specific objectives: 1) Develop and implement a preceptorship-based CME complemented by a web site for physicians and nurses working in Family Medicine Groups (FMGs). This CME will be based on needs assessment and will be validated by one FMG using questionnaires and semi structured interviews. Also, references and teaching tools will be available for participants on the web site. 2) Establish a collaborative intra/inter-regional interdisciplinary network to enable on-going expertise update and networking for FMG teams. This tool consists of a discussion forum including exchanges about difficult "cases" and a monthly virtual meeting of all participants. 3) Evaluate the implementation of this integrated system at the level of the ability to form a number of 8 FMGs/year, access and utilization of the electronic tools and participants' satisfaction (physicians, nurses and experts). This will be measured with the help of questionnaires and web logging tools. Questionnaires and group interviews will also be performed in order to evaluate participants' satisfaction. 4) Determine the impact for the participants at the level of knowledge and expertise, attitudes and perceptions, and self-efficacy regarding the management of obesity. Questionnaires and interviews will be used to this purpose. 5) Deliver transferable knowledge for health professionals and decision-makers. Strategies and pitfalls of setting up this program will be identified, performance indicators series will be developed and accessibility to care will be evaluated for each FMG and the 2nd line team. A knowledge transfer plan will be elaborated and applied.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals working in a Family Medicine Group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in attitudes toward obese individual at 1 year | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculté de médecine, Université de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Baillargeon JP, St-Cyr-Tribble D, Xhignesse M, Brown C, Carpentier AC, Fortin M, Grant A, Simoneau-Roy J, Langlois MF. Impact of an educational intervention combining clinical obesity preceptorship with electronic networking tools on primary care professionals: a prospective study. BMC Med Educ. 2020 Oct 14;20(1):361. doi: 10.1186/s12909-020-02248-5. PMID 33054845